CLINICAL TRIAL: NCT03404531
Title: Reaching Black/African American and Hispanic/Latino MSM Through Social Media About Treatment as Prevention and Pre-Exposure Prophylaxis
Brief Title: Project Minority AIDS Prevention: Reaching Black and Hispanic MSM About PrEP and TasP Using Social Media
Acronym: MAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brown University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jacob J. van den Berg, PhD, Assistant Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U01PS005117 (NIH)
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Media Messages Intervention Group (Experimental): Participants randomized to this condition will have access to a newly developed, culturally-tailored interactive website and theoretically-grounded social media messages.
  Interventions: Behavioral: Social Media Messages Intervention Group
- Website Only Group (Active Comparator): Participants randomized to this condition will have access to a newly developed, culturally-tailored interactive website only.
  Interventions: Behavioral: Website Only Group

INTERVENTIONS:
Behavioral: Social Media Messages Intervention Group — The Social Media Messages Intervention Group will receive theoretically-grounded messages through social media in order to encourage participants to regularly access the newly developed, culturally-tailored website that includes information about treatment as prevention and pre-exposure prophylaxis.
  Arms: Social Media Messages Intervention Group
Behavioral: Website Only Group — The Website Only group will have access to the newly developed, culturally-tailored website but will not receive social media messages.
  Arms: Website Only Group

SUMMARY:
This project has the potential to improve the implementation science of treatment as prevention and pre-exposure prophylaxis uptake as a public health strategy for reducing new HIV infections in the United States. The investigators will develop and pilot test an intervention that combines messages sent over social media plus a newly developed interactive website specifically developed by and for Black/African American and Hispanic/Latino MSM to encourage treatment as prevention and pre-exposure prophylaxis use. Findings from this research can guide policy guidelines and recommendations for treatment as prevention and pre-exposure prophylaxis uptake for high-risk groups.

DETAILED DESCRIPTION:
For this Minority AIDS Research Project, the investigators will develop and pilot test an intervention to improve the science of treatment as prevention and pre-exposure prophylaxis uptake as a public health strategy to decrease new HIV infections among Black/African American and Hispanic/Latino men who have sex with men. This project uses a 3-phase study design to address the proposed Specific Aims. First, the investigators will use focus groups to gather feedback on our existing interactive Men2MenRI website that was developed for and by predominately White men who have sex with men in Rhode Island that includes information on treatment as prevention and pre-exposure prophylaxis, as well as other health and wellness topics to make it more culturally-tailored to Black/African American and Hispanic/Latino MSM. Second, the investigators will use cognitive interviewing techniques to develop and assess the acceptability of Information-Motivation-Behavioral/Social Cognitive Theory-grounded social media message content designed to motivate and encourage access to a newly developed and culturally-tailored interactive website. Third, the investigators will pilot test a two-arm trial comparing the combination of sending Information-Motivation-Behavioral/Social Cognitive Theory-guided messages plus the newly developed and culturally-tailored interactive website (active arm) to the website alone (control arm) to examine whether the combination approach will: 1) increase treatment as prevention and pre-exposure prophylaxis uptake (primary outcome); 2) increase knowledge of, more favorable attitudes toward, and increase behavioral intentions of treatment as prevention and pre-exposure prophylaxis use behaviors (exploratory outcome). This study is innovative in the use of a combination approach to treatment as prevention and pre-exposure prophylaxis uptake that leverages advances in social media as a platform for motivating behavior change.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or older 2. Biological male 3. Black/African American or Hispanic/Latino 4. History of condomless receptive or insertive anal intercourse with other men in the past 6 months 5. Currently using or have access and willingness to use social media over the next 6 months 6. Self-identify as HIV-negative or HIV-positive at enrollment 7. Self-identify as not being on HIV treatment (antiretroviral therapy or pre-exposure prophylaxis) or in HIV care at enrollment 8. Able to give informed consent

-

Exclusion Criteria:

1. Individuals who are intoxicated
2. Individuals report being coerced to participate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2017-11-10 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
treatment as prevention and pre-exposure prophylaxis uptake | 6 months
  Participants uptake of treatment as prevention and pre-exposure prophylaxis

SECONDARY OUTCOMES:
treatment as prevention and pre-exposure prophylaxis knowledge, attitudes, and behavioral intentions | 6 months
  assessment of knowledge, attitudes, and behavioral intentions toward treatment as prevention and pre-exposure prophylaxis use

CONTACTS AND LOCATIONS:
Overall Officials: Jacob J van den Berg, PhD, Principal Investigator — Brown University
Locations (1):
- Center for Alcohol and Addiction Studies, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Research data will be shared openly, proactively, and timely in accordance with the most recent NIH guidelines (http://grants.nih.gov/grants/policy/data_sharing/) while being mindful that the confidentiality and privacy of participants in research must be protected at all times. Specific plans to share data, including an overview of what will be shared, when it will be shared, how it will be shared, and who will have access to the data will be proposed in a data sharing agreement that all investigators and prospective users of the data will complete when requesting access to the data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available to the public three years after study has been completed.
Access Criteria: Requests for data will be reviewed by the PI and persons who request data will be required to submit a proposal and to sign an agreement form.

REFERENCES:
- [Derived] van den Berg JJ, Silverman T, Fernandez MI, Henny KD, Gaul ZJ, Sutton MY, Operario D. Using eHealth to Reach Black and Hispanic Men Who Have Sex With Men Regarding Treatment as Prevention and Preexposure Prophylaxis: Protocol for a Small Randomized Controlled Trial. JMIR Res Protoc. 2018 Jul 16;7(7):e11047. doi: 10.2196/11047. PMID 30012549